CLINICAL TRIAL: NCT05534009
Title: Health Care Workers Cohort Study in the EuCARE Project (EuCARE-HCW)
Status: Recruiting | Type: Observational
Sponsor: Euresist Network GEIE (Other)
Collaborators: Centro Hospitalar Lisboa Ocidental (Other Government); ASST Santi Paolo e Carlo (Other); Bach Mai Hospital (Other); Hospital Regional de Alta Especialidad "Dr. Juan Graham Casasus" (Other); Heinrich-Heine University, Duesseldorf (Other); Istituto Europeo di Oncologia (Other); Vilnius University Hospital Santaros Klinikos (Other)
Responsible Party: Sponsor
Other Study IDs: EuCARE-HCW
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — biological material from healthcare workers from the Units partecipating
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Heath care workers (HCW): Adult (>18 years) HCW with mandatory information on their SARS-CoV-2 infection and vaccination status. For those with a history of SARS-CoV-2 infection, diagnosis obtained by detection of SARS-CoV-2 RNA
  Interventions: Other: Follow up of the first known immunization event

INTERVENTIONS:
Other: Follow up of the first known immunization event — The baseline for enrolment into the study is defined by the occurrence of the first known immunization event, either natural infection or vaccination. The follow-up is planned to last 24 months with respect to this baseline. In subjects with natural infection, the viral variant must be determined for each prospective case by analysis of a nasopharyngeal swab obtained as soon as possible at diagnosis. For historical cases where the variant was not determined and a contemporary nasopharyngeal swab has not been stored, the viral variant may be inferred when a specific variant was dominating the geographic area according to official records available at local health agencies. However, the variant assignment will be labelled as putative, rather than proved.
  HCWs can be enrolled in the category of:
  (i) vaccination not followed by any later infection, (ii) infection followed by vaccination and (iii) vaccination followed by infection.

SUMMARY:
The WP3 healthcare workers cohort in EuCARE is an observational multicentre study including collection of retrospective (historical) and prospective data and sample collection from health care workers with either a vaccination or a confirmed SARS-CoV-2 infection. Samples from HCW are sent to central laboratories for WP2 study were the impact of different variants in humoral and cellular immunity is to be analysed by biostatistical methods and with artificial intelligence in WP5. This analysis will focus on the impact on vaccine escape of viral variants / viral sequences as well as on any escape from any combination of natural and vaccine induced immunity. Eight countries will participate (Portugal, Italy, Germany, Lithuania, Georgia, Russia, Vietnam and Mexico).

DETAILED DESCRIPTION:
Background: Protection from SARS-CoV-2 infection is known to occur soon after vaccination or natural disease, fading over time. Although protection from serious illness does occur, protection from infection is insufficient and the impact of each variant and of each vaccine or vaccine schedule is a matter of continuous study. Recruiting participants from countries with different vaccines and vaccine schedules is of upmost importance to analyse these relationships and breakthrough infections. Study objectives: The EuCARE-HCW study contributes with data and samples from

HCW to EuCARE-IMMUNITY study that will analyse the NtAb and CMI to different SARS- CoV-2 variants following any combination of natural infection and vaccination. Specific

objectives include:

* to collect data and biological material from COVID-19 healthcare workers in 9 clinics from 8 countries and 3 continents.
* Enrolment of HCW with an immunogenic event, either vaccination or infection.
* Periodic collection of serum and whole blood every 4 months since enrolment and during 12-24 months (depending on how long immunity persists).
* Sample preparation, storage and shipment to central EuCARE laboratories where WP2 study group will analyse natural and artificial immunity to SARS-CoV-2 variants (EuCARE-IMMUNITY), namely:

  * Analyse the magnitude, breadth and duration of immunity following natural infection and/or vaccination.
  * Define the cross-immunity among the different viral variants.
  * Analyse the immune escape in a comprehensive set of combinations of vaccines and natural infection(s).
* To accomplish the above objectives, WP2 will test:

  * Neutralising antibodies
  * Cellular immunity
  * Viral sequences

ELIGIBILITY:
Inclusion Criteria:

The study subjects will be selected based on the following inclusion criteria:

1. Adult (>18 years) HCW with mandatory information on their SARS-CoV-2 infection and vaccination status.
2. For those with a history of SARS-CoV-2 infection, diagnosis obtained by detection of SARS-CoV-2 RNA
3. Having a signed informed consent when required by ethical approval

Exclusion Criteria: NONE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For each subject baseline will be the occurrence of the first known immunization event, either natural infection or vaccination. The follow-up is planned to last 24 months with respect to this baseline.
  Health CareWorkers can be enrolled in the category of:
  (i) vaccination not followed by any later infection, (ii) infection followed by vaccination and (iii) vaccination followed by infection. However, infections diagnosed during the first wave of the epidemic are suitable for the analysis of natural immunity to SARS-CoV-2 because vaccination was administered several months later.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of HCW involved in the study | through study completion, an average of 3 years
  To collect the higher possible number of data and biological materials from the HCWs of the participating Units

CONTACTS AND LOCATIONS:
Overall Officials: CRISTINA TOSCANO, DR, Study Chair — Centro Hospitalar de Lisboa Ocidental (CHLO)
Locations (7):
- Heinrich Heine university, Düsseldorf, Germany
- Italy (2):
  - Azienda Socio-Sanitaria Territoriale Santi Paolo e Carlo, Milan
  - Ieo Istituto Europeo Di Oncologia, Milan
- Viesoji Istaiga Vilniaus Uiversiteto Ligoninė Santaros klinikos, Vilnius, Lithuania
- Hospital Juan Ghaham Casasus, Villahermosa, Mexico
- Centro Hospitalar de Lisboa Ocidental, Lisbon, Portugal
- Bach Mai Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
The study is part of a project funded by the European Commission and the project agreement with theCommission affirms that the data and the results will be publi
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: AFTER THE STUDY END NO TIME LIMIT WAS FIXED
Access Criteria: REQUEST TO THE STUDY COORDINATOR OR TO THE PROJECTPARTNERS
URL: https://eucareresearch.eu/